CLINICAL TRIAL: NCT02022280
Title: Do Proton Pump Inhibitors (PPIs) Increase Cardiovascular Risk? Effect of PPIs on Endothelial Function and ADMA.
Brief Title: Effect of Proton Pump Inhibitors on Endothelial Function
Acronym: PPI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 23848; 1144447-121-DHAXB (Other Grant/Funding Number: Stanford Translational Research and Applied Medicine)
Record Dates: First submitted 2013-12-03; First posted 2013-12-27 (Estimated); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Endothelial Dysfunction
MeSH Terms: interventions — Lansoprazole

ARMS (2):
- Proton Pump Inhibitor (Experimental): Lansoprazole (Prevacid)
  Interventions: Drug: Lansoprazole
- Vitamin pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lansoprazole
  Other Names: Prevacid
  Arms: Proton Pump Inhibitor
Drug: Placebo — Vitamin pill
  Arms: Vitamin pill

SUMMARY:
In this randomized controlled crossover study, the investigators propose to test the hypothesis that proton pump inhibitors (PPIs) increase plasma levels of asymmetric dimethylarginine (ADMA), which is a marker of endothelial dysfunction. The authors propose to evaluate ADMA concentrations and vascular function analysis in healthy volunteers and adults with a history of cardiovascular disease given PPI vs placebo for four weeks each.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers aged 18 to 75 years (n=10) or male or female volunteers with a history of coronary or peripheral artery disease (n=10)
* Able to understand the nature of the study and to give written informed consent
* Able to communicate well with the investigator himself or his/her representatives
* Body Mass Index between 18 kg/m^2 and 35 kg/m^2 at the screening visit
* Creatinine <1.5, and liver enzymes <2x normal, with all laboratory tests considered normal or of no significant clinical relevance to the study by the investigator

Exclusion Criteria:

* Contra-indication to proton pump inhibitor treatment
* Current treatment with PPI or H2 antagonist, and not able to tolerate withdrawal or washout of medication.
* Current or historical evidence of clinically severe cardiovascular, neurological, hematological, hepatic, gastrointestinal, renal, pulmonary, endocrinological, metabolic or psychiatric disease.
* Any other acute or chronic disease which could influence the volunteer's health and/or the study results
* Presence or history of malabsorption or any gastrointestinal surgery except appendectomy or hernia repair
* Use of enzyme inducers or enzyme inhibitor drugs within the last three months before the first drug administration
* Participation in another ongoing clinical trial
* Past or current drug exposure amounting to drug abuse or addiction
* Past or current alcohol exposure amounting to alcohol abuse or addiction (i.e. > 28 units per week for males, where 1 unit = one measure of spirit (25 mL), one glass of wine (125 mL) or 1/2 pint beer)
* Donation of blood or any other major blood loss (>500 mL) within three months before the study
* Unwilling or unable to comply with the study protocol for any reason or in the opinion of the investigator should not participate in the study
* Positive test for hepatitis B surface antigen, hepatitis C antibody, HIV-1 or HIV-2 antibody at screening
* Known allergy or intolerance to any other compound in the study drug or any other closely related compound

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in reactive hyperemia index as measured by peripheral arterial tonometry (EndoPAT) | Baseline, 1 week, 5 weeks, 7 weeks, 11 weeks, 12 weeks

SECONDARY OUTCOMES:
Change in blood ADMA level | Baseline, 1 week, 5 weeks, 7 weeks, 11 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Leeper, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- [Result] Ghebremariam YT, Cooke JP, Khan F, Thakker RN, Chang P, Shah NH, Nead KT, Leeper NJ. Proton pump inhibitors and vascular function: A prospective cross-over pilot study. Vasc Med. 2015 Aug;20(4):309-16. doi: 10.1177/1358863X14568444. Epub 2015 Apr 2. PMID 25835348